CLINICAL TRIAL: NCT04191018
Title: Progression of Gastroesophageal Varices After Sustained Virological Response by Interferon-free Regimens in Patients With Advanced Fibrosis / Cirrhosis Due to Chronic Hepatitis C
Brief Title: GastrOesophageal Varices After Sustained Virological Response
Acronym: GOVaSViR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oswaldo Cruz Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 10320319.6.0000.5262
Record Dates: First submitted 2019-11-27; First posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Liver Diseases; Hepatitis C
Keywords: sustained virological response; portal hypertension; cirrhosis; gastrointestinal endoscopy
MeSH Terms: conditions — Liver Diseases; Hepatitis C; Hypertension, Portal; Fibrosis | interventions — Endoscopy, Gastrointestinal; Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Liver elastography — Liver stiffness measurement
  Other Names: transient elastography (Fibroscan); 2D-shear wave (GE Healthcare); point-shear wave (Phillips)
Diagnostic Test: Splenic elastography — Splenic stiffness measurement
  Other Names: transient elastography (Fibroscan); 2D-shear wave (GE Healthcare); point-shear wave (Phllips)
Diagnostic Test: Gastrointestinal endoscopy — Gastrointestinal endoscopy
  Other Names: esophagogastroduodenoscopy

SUMMARY:
Chronic hepatitis C remains a public health issue because up to 70 million people are chronically infected by hepatitis C virus (HCV) worldwide. Presence of advanced fibrosis/cirrhosis might be associated with liver-related complications, such as hepatocellular carcinoma and oesophageal varices bleeding. Oesophageal varices (OV) might be present in up to 40% of patients with liver cirrhosis have and the mortality rates from bleeding might be up to 20% per episode. Early diagnosis of advanced fibrosis/cirrhosis associated with hepatitis C treatment are key features for preventive and therapeutic measures to reduce liver-related mortality in HCV-infected patients.

Liver elastography is a high accurate non-invasive test for diagnosis of advanced fibrosis/cirrhosis. Few different methods of liver elastography are currently available: transient elastography by Fibroscan and ultrasound elastography by point-shear wave (p-SWE) and 2D-shear wave (2D-SWE). Gastrointestinal endoscopy (GIE) has been considered the gold standard for screening or surveillance of esophageal varices. More recently, international guidelines have been recommending the use of non-invasive methods to indicate or avoid OV screening: Baveno VI guidelines proposed that compensated cirrhotic patients with a liver stiffness measurement (LSM) by transient elastography <20kPa and a platelet count >150,000/μL can avoid screening endoscopy. The use of direct-acting agents (DAAs) has revolutionized the treatment of chronic hepatitis C with high effectiveness shown using all-oral interferon-free regimens. HCV cure, sustained virological response (SVR), has been associated with lower rates of liver-related complications, increase in quality of life and decrease in waiting-list registrations for liver transplantation in patients with chronic hepatitis C. Preliminary studies have been reporting significant regression liver stiffness after SVR. However, it is unclear whether SVR might decrease portal hypertension leading to OV regression and a reduced risk of variceal bleeding. In addition, the use of non-invasive methods to avoid OV screening must be validated in HCV patients after SVR. The aims of this cross-sectional study with prospective inclusion of patients will be: (i) to evaluate the impact of SVR in portal hypertension in HCV patients with advanced fibrosis/liver cirrhosis treated by interferon-free regimens and (ii) to validate non-invasive methods to avoid OV screening by GIE

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Presence of advanced fibrosis or cirrhosis (stage F≥3 METAVIR) based on liver stiffness by transient elastography (≥ 9,5 kPa) or liver biopsy
* Gastrointestinal endoscopy at least 24 months before start of direct-acting agents for HCV treatment
* Liver stiffness measurement at least 18 months after SVR

Exclusion Criteria:

* Autoimmune hepatitis, hepatosplenic schistosomiasis or cholestasis diseases
* Liver transplantation
* Presence of high volume ascites or hepatocellular carcinoma
* Participation in programs of esophageal band ligation for eradication of esophageal varices
* Presence of signs of acute decompensated liver disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced fibrosis or cirrhosis with sustained virologic response by direct-acting agents for HCV treatment
Sampling Method: Non-Probability Sample
Enrollment: 322 (Estimated)
Dates: Start 2019-11-26 (Estimated); Primary Completion 2022-08-14 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of esophageal varices (portal hypertension) after SVR | up to 48 months after SVR
  Evaluation of presence/absence of esophageal varices after SVR in patients with advanced fibrosis or cirrhosis compared to before treatment
Validation of the Baveno's criteria to avoid gastrointestinal endoscopy for screening of esophageal varices after SVR | up to 48 months after SVR
  Validation of the diagnostic performance of non-invasive tests (liver and splenic stiffness or biological markers) to screen esophageal varices in patients with advanced fibrosis/cirrhosis after SVR by DAA treatment for HCV

SECONDARY OUTCOMES:
Incidence of regression of esophageal varices after SVR | up to 48 months after SVR
  Evaluation of absence of esophageal varices after SVR in patients with advanced fibrosis or cirrhosis and esophageal varices before treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Perazzo, PhD, Principal Investigator — Oswaldo Cruz Foundation
Locations (2):
- Brazil (2):
  - Evandro Chagas National Institute of Infectious Diseases, Rio de Janeiro, Rio de Janeiro/RJ
  - Bonsucesso Federal Hospital, Rio de Janeiro